CLINICAL TRIAL: NCT05155787
Title: Construction and Evaluation of Neurofeedback Training (NFT) on Sleep Quality and Cognitive Function Performance Among HIV-infected Persons
Brief Title: Neurofeedback Training (NFT) on Sleep Quality and Cognitive Function Performance Among HIV-infected Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-BR-109-031
Record Dates: First submitted 2021-04-04; First posted 2021-12-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-07

CONDITIONS: Poor Quality Sleep; HIV Infections
Keywords: neurocognitive performance, neurofeedback training
MeSH Terms: conditions — HIV Infections | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with neurofeedback training (Experimental): The neurofeedback training system records the brain waves from the subject and converts the original brain wave signal into frequency energy through spectrum analysis. The system will help the subject to find self relax method for producing more alpha waves. Each person will arrange training three times a week for four weeks.
  Interventions: Device: Neurofeedback
- Group with shame neurofeedback training (Sham Comparator): In the shame group, the system is not feedback to the actual wave. Each person will arrange training three times a week for four weeks.
  Interventions: Device: Shame neurofeedback

INTERVENTIONS:
Device: Neurofeedback — Neurofeedback training as a method is going to let the brain producing the alpha signal (8-13 Hz).
  Arms: Group with neurofeedback training
Device: Shame neurofeedback — shame neurofeedback
  Arms: Group with shame neurofeedback training

SUMMARY:
The purpose of this study is to evaluate the effects of NFT on sleep quality and cognitive-behavioral performance among HIV-infected patients, to use it as a reference for the construction of NFT as a clinical empirical treatment model for HIV-infected patients with sleep disturbance.

DETAILED DESCRIPTION:
This study will aim to evaluate the effects of NFT on sleep quality and neurocognitive performance among HIV-infected persons with sleep disturbance. A double-blind clinical randomized parallel trial will be enrolled in HIV-infected persons with sleep disturbance. We will exclude subjects with OSA. Random sampling by using a computer, and then we will be divided subjects into 2 groups. 30 people will be drawn into the experimental group and control group (sham). Two groups will be treated with NFT three times a week for at least four weeks. The vague distribution of this study will be handled by SNOSE (Sequentially Numbered, Opaque, Sealed Envelopes). Double-blind subjects include subjects, family members, outcome appraisers, and technologists to ensure the integrity of randomized controlled trials and blind assignment. The outcome indicators are sleep quality and the Chinese Montreal cognitive assessment (MoCA). Treatment compliance, sample loss, and adverse event events will be monitored, and the analysis will be followed the principle of intention to treat. The pair student t or McNemar's test will use to test the effect of NFT on sleep quality and neurocognitive performances among HIV-infected persons.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected persons

Exclusion Criteria:

* Patients with central neural infections
* Pregnant women
* Drug or alcohol abuse

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality as assessed by Chinese version Pittsburgh Sleep Quality Index (CPSQI) | 1 month
  Subjective sleep quality was measured by Chinese version of the Pittsburgh Sleep Quality Index (CPSQI). A patient with a score of >=5 would be identified as poor sleep quality.
The length of minutes of total sleep time (TST) as assessed by the acti-watch | 1 month
  This objective outcome measures by the acti-watch (Axivity, Newcastle, UK), which contains an accelerometer for detection of movement, produces a continuous electrical signal (voltage) when a participant wore the device for up to one month.
  Total sleep time (TST): TST referred to as the true sleep period, is defined as the interval (within time in bed) from sleep onset to sleep offset.
The length of minutes of sleep onset latency (SOL) as assessed by the acti-watch | 1 month
  This objective outcome measures by the acti-watch (Axivity, Newcastle, UK), which contains an accelerometer for detection of movement, produces a continuous electrical signal (voltage) when a participant wore the device.
  Sleep onset latency (SOL): SOL refers to the number of minutes it took a subject to fall asleep. It is the number of minutes between lying down in bed and actually falling asleep.
The percentage of sleep efficiency (SE) as assessed by the acti-watch | 1 month
  This objective outcome measures by the acti-watch (Axivity, Newcastle, UK), which contains an accelerometer for detection of movement, produces a continuous electrical signal (voltage) when a participant wore the device for up to one month.
  Sleep efficiency (SE): SE is defined as the percentage of time spent asleep during the time in bed. SE is derived as follows: SE=(TST/time in bed)×100%.

SECONDARY OUTCOMES:
Cognitive performance as assessed by the International HIV dementia scale (IHDS) | 1 month
  We will evaluate cognitive performance using International HIV dementia scale (IHDS). The maximum possible score is 12 points. A patient with a score of ≤10 should be evaluated further for possible HIV dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alford K, Banerjee S, Nixon E, O'Brien C, Pounds O, Butler A, Elphick C, Henshaw P, Anderson S, Vera JH. Assessment and Management of HIV-Associated Cognitive Impairment: Experience from a Multidisciplinary Memory Service for People Living with HIV. Brain Sci. 2019 Feb 8;9(2):37. doi: 10.3390/brainsci9020037. PMID 30744034
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Gamaldo CE, Gamaldo A, Creighton J, Salas RE, Selnes OA, David PM, Mbeo G, Parker BS, Brown A, McArthur JC, Smith MT. Evaluating sleep and cognition in HIV. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):609-16. doi: 10.1097/QAI.0b013e31829d63ab. PMID 23722610